CLINICAL TRIAL: NCT05177432
Title: Quadratic Phenotypic Optimisation Platform (QPOP) Utilisation to Enhance Selection of Patient Therapy Through Patient Derived Organoids in Breast Cancer
Acronym: QUEST
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BR02/03/21
Record Dates: First submitted 2021-11-10; First posted 2022-01-04 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
Keywords: QPOP; Enhance Selection; Patient Therapy; Patient Derived Organoids; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-centre study based on the Simon 2-stage optimal design: 9 patients will be enrolled initially. The study will be expanded to a further 14 patients (Stage II) if 2 or more patients enrolled in stage I of the study achieve an objective response (of >35% ) with the chemotherapeutic agent selected by the drug screen assay. Accounting for 10% attrition rate, a total of 26 evaluable patients will be included in both stages of study.
  QPOP-based drug screen assay will be used as a clinical decision platform to identify patient-specific drug combinations across a range of breast cancer patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QPOP-based drug screen assay using patient tumour-derived organoids (Experimental): Patients with Histological confirmed breast carcinoma of any subtype (any estrogen receptor, progesterone receptor and HER2 receptor status) with at least 1 tumour lesion (primary or metastatic) amendable to fresh biopsy and measurable based on RECIST 1.1 criteria will undergo biopsy to obtain a sample of cancer tissue that will be used to generate Patient Derived Organoids (PDOs).
  Patients' cells will be subjected to testing with 10-12 anti-cancer drugs and a table for treatment sensitivity to each drug will be derived after 8 to 12 weeks of treatment in the laboratory. Results will be reviewed at an expert panel discussion to decide on the most suitable anti-cancer drug treatment
  Interventions: Device: QPOP

INTERVENTIONS:
Device: QPOP — QPOP will be used as a clinical decision support platform to identity suitable patient-specific drug combinations across a range of breast cancer patients, which are derived from drug sensitivity tests using patient-derived materials.

SUMMARY:
Based on proof-of-concept study, the investigators hypothesise that the QPOP prediction model can be further extended into use in solid tumors. Using breast cancer as a model, the investigators intend to investigate the feasibility of QPOP as a clinical decision support platform to identify patient-specific drug combinations across a range of breast cancer patients. The investigators propose a pilot phase I clinical study to test the feasibility of using QPOP to guide therapy in patients with advanced breast cancer.

DETAILED DESCRIPTION:
Breast cancer (BC) is highly heterogeneous with more than 20 genetically, morphologically and clinically distinct subtypes. Despite improved diagnosis and a wide repertoire of clinically-approved therapies, metastatic BC patients have a dismal 5-year survival rate of about 20%. Systemic treatment options for breast cancer are empiric based on large clinical studies, and the ability to tailor choices individualized to each patient may aid optimization of patient's responses to treatment.

A major obstacle for drug development is the lack of clinically relevant cell model systems. The use of conventional two-dimensional (2D) cell cultures presents limitations in the recapitulation of the primary disease characteristics. In particular, monolayer cultures have been demonstrated for not being able to recapitulate the heterogeneous nature of primary patient tumor tissues. Despite the establishment of the National Cancer Institute 60 Panel (NCI-60) in an attempt to capture the heterogeneous nature of nine different cancer types, it is still unable to comprehensively represent the diversity which cancer patients exhibit, and is currently being phased out. Studies comparing the molecular profiles of cell lines with primary tumors have reported that conventional cell lines are unable to represent all cancer subtypes. Recently, patient-derived organoids (PDOs) has been demonstrated to faithfully preserve and maintain heterogeneity of several primary cancer types including BC and are being used to evaluate drug sensitivity and their associated genomic variations. PDOs have also been shown to retain the molecular profiles of the parental tumors and can be effectively used to investigate drug responses and mechanisms ex vivo. Thus, human PDOs can provide more clinically relevant models that can recapitulate disease heterogeneity for more accurate studies of drug responses as compared to conventional cell line-based models.

Identifying the most suitable patient-specific drug combinations remains a challenge due to the complex molecular networks that contribute to feedback mechanisms of drug resistance and compensatory oncogenic drivers that limit efficacy of targeted inhibitors. Pharmacogenomics is highly useful in predicting drug sensitivity and clinical outcome and define appropriate subpopulations for specific drugs based on genetic biomarkers. These approaches are largely limited to monotherapy and cannot identify patient-specific drug combinations nor do they consider other genomic alterations that are unaccounted for by the specific biomarkers used. In order to address this critical deficit in combination therapy, the investigators have developed an experimental-analytical hybrid platform, Quadratic Phenotypic Optimisation Platform (QPOP), that can rank potential drug combination response in biological model systems. The investigators initially applied QPOP towards identifying novel drug combinations against bortezomib-resistant multiple myeloma. As the investigators have improved the efficiency of the QPOP platform and applied QPOP towards primary patient samples and patient-derived organoids, it has become clear that QPOP may be useful as a clinical decision support platform that may be able to suggest clinically actionable and suitable patient-specific drug combinations derived from drug sensitivity tests using patient-derived materials.

The investigators hypothesise that the QPOP prediction model can be further extended into use in solid tumors. Using breast cancer as a model, we intend to investigate the feasibility of QPOP as a clinical decision support platform to identity patient-specific drug combinations across a range of breast cancer patients. The Investigators propose a pilot phase I clinical study to test the feasibility of using QPOP to guide therapy in patients with advanced breast cancer.

Eligible patients will undergo a fresh biopsy of tumour lesion to obtain cells that will be used to generate patient-derived tumour organoids. After successful organoid generation, organoids will be subjected to a 12-drug panel screening including 10 fixed drugs and 2 drugs that may be selected by physician based on treatment history of individual patients. The drug panel is curated taking into account standard drugs commonly used in breast cancer treatment as well as drugs/combinations being tested at ongoing therapeutic trials at the National University Cancer Institute Singapore (NCIS) which enrolled patients can gain access to. Fixed drug panel will include chemotherapy (cisplatin, 5-fluorouracil, paclitaxel), endocrine therapy (tamoxifen, fulvestrant), HER2-directed therapy (lapatinib) and small molecule tyrosine kinase inhibitors (abemaciclib, olaparib, alpelisib, lenvatinib).

QPOP analysis results will be reported to treating physician once available to aid selection of therapy. To prevent delay in patient treatment while awaiting QPOP results, patients are allowed to receive next line of therapy at physician's discretion (termed "empirical therapy"), and QPOP analyses results can be used to guide further lines of treatment upon progression on "empirical therapy".

ELIGIBILITY:
Part A - Inclusion and exclusion criteria to be fulfilled both prior to study enrolment and prior to commencement of study drug

Inclusion Criteria:

* Age >= 21 years.
* Histological confirmed breast carcinoma of any subtype (any estrogen receptor, progesterone receptor and HER2 receptor status)
* ECOG 0-1.
* At least 1 tumour lesion (primary or metastatic) amenable to fresh biopsy
* At least 1 measurable tumour lesions based on RECIST 1.1 criteria
* Estimated life expectancy of at least 12 weeks.
* Has documented progressive disease from last line of therapy.
* Has received at least 1 line of palliative systemic therapy
* Expected adequate organ function (bone marrow, hepatic, renal) after recovering from treatment-induced acute toxicities at the time of study treatment.
* Signed informed consent from patient or legal representative.
* Able to comply with study-related procedures.

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons:

* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Active bleeding disorder or bleeding site.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* History of significant neurological or mental disorder, including seizures or dementia.

Part B - Additional inclusion and exclusion criteria to be fulfilled prior to commencement of study drug

Inclusion criteria

Patients may be included in the study only if they meet all of the following criteria:

• Adequate organ function including the following:

Bone marrow:

* Absolute neutrophil (segmented and bands) count (ANC) >= 1.5 x 109/L
* Platelets >= 100 x 109/L
* Hemoglobin >= 8 x 109/L

Hepatic:

* Bilirubin <= 1.5 x upper limit of normal (ULN),
* ALT or AST <= 2.5x ULN, (or <=5 X with liver metastases)

Renal:

- Creatinine <= 1.5x ULN

Exclusion criteria

Patients will be excluded from the study for any of the following reasons:

* Treatment within the last 30 days with any investigational drug.
* Concurrent administration of any other tumour therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy at time of commencement of study drug.
* Major surgery within 28 days of study drug administration.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Non-healing wound.
* Poorly controlled diabetes mellitus.
* Symptomatic brain metastasis.
* Contraindication to receiving specific QPOP-directed study treatment within drug that has been recommended based on QPOP analyses (e.g., poorly controlled diabetes mellitus for alpelisib, left ventricular ejection fraction of <50% for trastuzumab-emtansine)
* Received more than 2 lines of empirical therapy between tumor biopsy for organoids growth and commencement on QPOP-directed study treatment (including endocrine therapy, chemotherapy, targeted therapy or immunotherapy)
* Biopsy for organoids growth performed more than 12 months from time of study drug commencement
* Has not recovered from acute toxicities from prior anti-cancer therapy

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer study - 99.9% breast cancer patients are female. Male breast cancer is extremely rare and we do not intend to include this rare population
Enrollment: 26 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2025-01-03 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate measured by RECIST 1.1 criteria to anti-cancer therapy selected by QPOP (prospective analysis). | 3 years

SECONDARY OUTCOMES:
Clinical benefit rate as determined by proportion of patients with complete response, partial response or stable disease as best response on RECIST 1.1 criteria (prospective analysis) | 3 years
Progression-free survival of QPOP-guided therapy as measured by RECIST 1.1 criteria (prospective analysis) | 3 years
Correlating QPOP prediction score of immediate past line of therapy and objective response rate to that therapy (retrospective correlative analysis) | 3 years
Correlating objective response rate (ORR) measured by RECIST v1.1 of the tumor lesion biopsied for QPOP analyses with QPOP guided therapy (retrospective correlative analysis) | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Fong ELS, Toh TB, Yu H, Chow EK. 3D Culture as a Clinically Relevant Model for Personalized Medicine. SLAS Technol. 2017 Jun;22(3):245-253. doi: 10.1177/2472630317697251. Epub 2017 Mar 9. PMID 28277923
- [Result] Gillet JP, Varma S, Gottesman MM. The clinical relevance of cancer cell lines. J Natl Cancer Inst. 2013 Apr 3;105(7):452-8. doi: 10.1093/jnci/djt007. Epub 2013 Feb 21. PMID 23434901
- [Result] Ledford H. US cancer institute to overhaul tumour cell lines. Nature. 2016 Feb 25;530(7591):391. doi: 10.1038/nature.2016.19364. No abstract available. PMID 26911756
- [Result] Virtanen C, Ishikawa Y, Honjoh D, Kimura M, Shimane M, Miyoshi T, Nomura H, Jones MH. Integrated classification of lung tumors and cell lines by expression profiling. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12357-62. doi: 10.1073/pnas.192240599. Epub 2002 Sep 6. PMID 12218176
- [Result] Goodspeed A, Heiser LM, Gray JW, Costello JC. Tumor-Derived Cell Lines as Molecular Models of Cancer Pharmacogenomics. Mol Cancer Res. 2016 Jan;14(1):3-13. doi: 10.1158/1541-7786.MCR-15-0189. Epub 2015 Aug 6. PMID 26248648
- [Result] Sachs N, de Ligt J, Kopper O, Gogola E, Bounova G, Weeber F, Balgobind AV, Wind K, Gracanin A, Begthel H, Korving J, van Boxtel R, Duarte AA, Lelieveld D, van Hoeck A, Ernst RF, Blokzijl F, Nijman IJ, Hoogstraat M, van de Ven M, Egan DA, Zinzalla V, Moll J, Boj SF, Voest EE, Wessels L, van Diest PJ, Rottenberg S, Vries RGJ, Cuppen E, Clevers H. A Living Biobank of Breast Cancer Organoids Captures Disease Heterogeneity. Cell. 2018 Jan 11;172(1-2):373-386.e10. doi: 10.1016/j.cell.2017.11.010. Epub 2017 Dec 7. PMID 29224780
- [Result] Vlachogiannis G, Hedayat S, Vatsiou A, Jamin Y, Fernandez-Mateos J, Khan K, Lampis A, Eason K, Huntingford I, Burke R, Rata M, Koh DM, Tunariu N, Collins D, Hulkki-Wilson S, Ragulan C, Spiteri I, Moorcraft SY, Chau I, Rao S, Watkins D, Fotiadis N, Bali M, Darvish-Damavandi M, Lote H, Eltahir Z, Smyth EC, Begum R, Clarke PA, Hahne JC, Dowsett M, de Bono J, Workman P, Sadanandam A, Fassan M, Sansom OJ, Eccles S, Starling N, Braconi C, Sottoriva A, Robinson SP, Cunningham D, Valeri N. Patient-derived organoids model treatment response of metastatic gastrointestinal cancers. Science. 2018 Feb 23;359(6378):920-926. doi: 10.1126/science.aao2774. PMID 29472484
- [Result] Shaughnessy JD Jr, Qu P, Usmani S, Heuck CJ, Zhang Q, Zhou Y, Tian E, Hanamura I, van Rhee F, Anaissie E, Epstein J, Nair B, Stephens O, Williams R, Waheed S, Alsayed Y, Crowley J, Barlogie B. Pharmacogenomics of bortezomib test-dosing identifies hyperexpression of proteasome genes, especially PSMD4, as novel high-risk feature in myeloma treated with Total Therapy 3. Blood. 2011 Sep 29;118(13):3512-24. doi: 10.1182/blood-2010-12-328252. Epub 2011 May 31. PMID 21628408
- [Result] Rashid MBMA, Toh TB, Hooi L, Silva A, Zhang Y, Tan PF, Teh AL, Karnani N, Jha S, Ho CM, Chng WJ, Ho D, Chow EK. Optimizing drug combinations against multiple myeloma using a quadratic phenotypic optimization platform (QPOP). Sci Transl Med. 2018 Aug 8;10(453):eaan0941. doi: 10.1126/scitranslmed.aan0941. PMID 30089632
- [Result] de Mel S, Rashid MBM, Zhang XY, Goh J, Lee CT, Poon LM, Chan EHL, Liu X, Chng WJ, Chee YL, Lee J, Yuen YC, Lim JQ, Chia BKH, Laurensia Y, Huang D, Pang WL, Cheah DMZ, Wong EKY, Ong CK, Tang T, Lim ST, Ng SB, Tan SY, Loi HY, Tan LK, Chow EK, Jeyasekharan AD. Application of an ex-vivo drug sensitivity platform towards achieving complete remission in a refractory T-cell lymphoma. Blood Cancer J. 2020 Jan 27;10(1):9. doi: 10.1038/s41408-020-0276-7. No abstract available. PMID 31988286